CLINICAL TRIAL: NCT00595114
Title: Ancillary Study of Oxidative Stress and Anti-Inflammatory Lipids in Airway Disease in the MIA (ACRN) and LEUKO (CCRN) Trials
Brief Title: Association Between Increased Oxidative Stress, Anti-Inflammatory Fatty Acid Formation, and Airway Infection in People With Asthma and Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce D. Levy, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 1421; R01HL090927 (NIH); HL090927
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Airway; Inflammation; Infection; Lipid Mediators; Oxidative Stress
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Inflammation; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and sputum samples with DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- MIA 1: Participants from the MIA trial who are polymerase chain reaction (PCR) negative and have received treatment with placebo
- MIA 2: Participants from the MIA trial who are PCR negative and have received treatment with the antibiotic clarithromycin
- MIA 3: Participants from the MIA trial who are PCR positive and have received treatment with placebo
- MIA 4: Participants from the MIA trial who are PCR positive and have received treatment with the antibiotic clarithromycin
- LEUKO 1: Participants from the LEUKO trial who have received treatment with placebo
- LEUKO 2: Participants from the LEUKO trial who have received treatment with zileuton

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and asthma are common respiratory diseases in which people experience long-term inflammation of the lungs. Exacerbations, or prolonged worsening of symptoms, of asthma and COPD are often life-threatening and can lead to frequent need for hospitalization. Even with the proper use of bronchodilators, corticosteroids, and other currently available medications, clinical responses among people with COPD and asthma are variable. There remains a significant unmet clinical need for new therapeutic approaches and insights, including the identification of biomarkers to accurately assess the presence of airway infection and intensity of airway inflammation. This study will investigate potential natural biological causes and new biomarkers for increased susceptibility to persistent airway infection in asthma and COPD.

DETAILED DESCRIPTION:
COPD and asthma are chronic lung diseases that result in impaired air flow in the lungs, often causing coughing, wheezing, and shortness of breath. In uncontrolled COPD and asthma, people may experience a rapid worsening of symptoms, which may include fever, difficulty breathing, and chest pain. These exacerbations are the most serious expression of asthma and COPD and are usually caused by lung infections or air allergens. However, the biological basis for susceptibility to airway infection and inflammation is not well understood. Increased oxidative stress within the airways has been linked to several airway diseases. This increase in oxidative stress may reduce production of key fatty acid anti-inflammatory mediators. In turn, this may disrupt the airway's natural immune response mechanisms, making the airways more vulnerable to infection or inflammation during COPD and asthma exacerbations. This ancillary study will determine whether susceptibility to persistent airway infection in asthma and COPD stems from increased oxidative stress that impairs the natural formation of protective fatty acid mediators.

This ancillary study will use data biological samples, including blood and sputum, from participants currently enrolled in the Macrolides in Asthma (MIA; NCT00318708) and the Antileukotriene Therapy for COPD Exacerbations (KIA; NCT01097694). Biological samples will undergo fatty acid mediator analysis and RNA isolation. There will be no study visits for this study.

ELIGIBILITY:
Inclusion Criteria:

* No change from the MIA and LEUKO trials

Exclusion Criteria:

* No change from the MIA and LEUKO trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This ancillary study will use data and specimens previously collected in the Macrolides in Asthma (MIA) and the Antileukotriene Therapy for COPD Exacerbations (LEUKO) trials.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D. Levy, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ono E, Dutile S, Kazani S, Wechsler ME, Yang J, Hammock BD, Douda DN, Tabet Y, Khaddaj-Mallat R, Sirois M, Sirois C, Rizcallah E, Rousseau E, Martin R, Sutherland ER, Castro M, Jarjour NN, Israel E, Levy BD; National Heart, Lung, and Blood Institute's Asthma Clinical Research Network. Lipoxin generation is related to soluble epoxide hydrolase activity in severe asthma. Am J Respir Crit Care Med. 2014 Oct 15;190(8):886-97. doi: 10.1164/rccm.201403-0544OC. PMID 25162465

RESULTS

PARTICIPANT FLOW:
Groups:
- MIA 1: Participants from the MIA trial with mild asthma
- KIA 1: Participants from the KIA trial with severe asthma
Period: Overall Study
Arm/Group | MIA 1 | KIA 1
Started | 24 | 19
Completed | 24 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MIA 1 | KIA 1 | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10) | 40 (11) | 38 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 8 | 23
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 19 | 43

OUTCOME MEASURES:

1. Primary Outcome: 8-isoprostane Levels as Biochemical Markers for Nonenzymatic Oxidative Stress in Asthma
Description: 8-isoprostane levels in sputum
Time Frame: Measured at completion of sample analysis
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MIA 1 | KIA 1
Number analyzed (Participants) | 24 | 19
pg/ml | 292.4 (51.0) | 421.8 (195.4)

ADVERSE EVENTS:
Arm/Group | MIA 1 | KIA 1
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/19
Other Adverse Events (participants affected / at risk) | 0/24 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No